CLINICAL TRIAL: NCT02091050
Title: Clinical and Dosimetric Comparison of 2D Versus 3D HDR Brachytherapy
Brief Title: 2D vs 3D Planning for High-Dose Rate (HDR) Gynecological Brachytherapy
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: AC Camargo Cancer Center (Other)
Responsible Party: Principal Investigator, Lucas Gomes Sapienza, MD, AC Camargo Cancer Center
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: AC-G 01
Record Dates: First submitted 2014-03-13; First posted 2014-03-19 (Estimated); Last update posted 2018-08-31 (Actual); Status verified 2018-08

CONDITIONS: Cervix Cancer; Endometrial Cancer
Keywords: 3D Brachytherapy; cervical cancer; endometrial cancer; vaginal vault brachytherapy
MeSH Terms: conditions — Uterine Cervical Neoplasms; Endometrial Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- HDR Brachytherapy 24Gy (4 x 6Gy) (Other): Vaginal vault brachytherapy, associated or not with external beam radiotherapy.
  Interventions: Other: 2D HDR planning; Other: 3D HDR planning

INTERVENTIONS:
Other: 2D HDR planning — HDR planning using simple radiograph (2D)
Other: 3D HDR planning — HDR planning using computed tomography (3D)

SUMMARY:
Demonstrate the limitations of conventional dosimetry (2D) for the adjuvant brachytherapy treatment and assess whether tridimensional dosimetry relates more faithfully with the occurrence of adverse effects.

DETAILED DESCRIPTION:
Radiotherapy is part of a multidisciplinary strategy to fight cancer in all stages, using ionizing radiation to cause damage in tumor cells. After radical surgical treatment of gynecological tumors, pathological findings, such as extension of the myometrium invasion, histologic grade, and vascular- lymphatic invasion predict the risk of locoregional recurrence of disease and, consequently, the need for adjuvant treatment. There are two main methods of adjuvant therapy after hysterectomy for malignant neoplasm of the cervix or endometrium: external beam radiotherapy with or without booster dose of vaginal vault brachytherapy or brachytherapy alone. There are few data in the literature and clinical experience with brachytherapy dimensional (3D) for adjuvant treatment of vaginal vault .

Objective: To demonstrate the limitations of conventional dosimetry (2D) for the adjuvant brachytherapy treatment and assess whether tridimensional dosimetry relates more faithfully with the occurrence of adverse effect.

Methods: A prospective study in the Department of Radiation Oncology, Antonio Candido Camargo Cancer Center will be developed with an expected duration of 14 months and will include 60 patients. Dosimetric parameters of brachytherapy treatment of vaginal vault, able to influence the incidence of adverse effects will be evaluated. Computed tomography for planning of external beam radiotherapy and brachytherapy planning will be used, after placement of intra- vaginal applicator and urinary catheter. For planning brachytherapy two fast acquisition sequences, one with a urinary catheter not pulled and pulled another with the probe will be obtained. The prescription dose obey the standard indication of document of the International Commission on Radiation Units & Measurements (ICRU 38).

ELIGIBILITY:
Inclusion Criteria:

* Malignant neoplasm of the cervix or endometrium;
* Tomography scan available in the planning system.

Exclusion Criteria:

* Patients did not undergo surgery as initial treatment;
* Patients without available tomography for planning;

Ages: 18 Years to 85 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2014-06; Primary Completion 2015-03 (Actual); Study Completion 2017-01 (Actual)

PRIMARY OUTCOMES:
Dosimetry of Organs of genitourinary and gastrointestinal tracts | one week after the tomograph
  Dose in bladder; rectum; small intestine; sigmoid colon; urethra; dose trigone; vaginal cuff.

SECONDARY OUTCOMES:
Cost analysis with local care. | 6 weeks
Acute Genitourinary Toxicity | 6 weeks
  toxicity associated with the genitourinary tract, using Common Terminology Criteria for Adverse Events v4.0 (CTCAE v4.0)
Acute Gastrointestinal toxicity | 6 weeks
  toxicity associated with the gastrointestinal tract, using Common Terminology Criteria for Adverse Events v4.0 (CTCAE v4.0)
Late Genitourinary Toxicity | 3 Years
  toxicity associated with the genitourinary tract, using Common Terminology Criteria for Adverse Events v4.0 (CTCAE v4.0)
Late Gastrointestinal toxicity | 3 Years
  toxicity associated with the gastrointestinal tract, using Common Terminology Criteria for Adverse Events v4.0 (CTCAE v4.0)

CONTACTS AND LOCATIONS:
Locations (1):
- AC Camargo Cancer Center, São Paulo, São Paulo, Brazil

REFERENCES:
- [Result] Sapienza LG, Flosi A, Aiza A, de Assis Pellizzon AC, Chojniak R, Baiocchi G. Volumetric (3D) bladder dose parameters are more reproducible than point (2D) dose parameters in vaginal vault high-dose-rate brachytherapy. Sci Rep. 2016 Jun 14;6:28074. doi: 10.1038/srep28074. PMID 27296459
- See also: Related Info — https://www.ncbi.nlm.nih.gov/pubmed/27296459